CLINICAL TRIAL: NCT06792279
Title: Use of Ultrasound Echo Intensity for the Detection of Muscle Quality in Children - Protocol for a Validation Study
Brief Title: Detection of Muscle Quality in Children - Protocol for a Validation Study
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Michal Šteffl, ass. prof., Charles University, Czech Republic
Other Study IDs: EK 101/2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the validity and reliability of ultrasound echo intensity (EI) as a diagnostic tool for assessing muscle quality in children aged 10-14 years, including normal-weight, obese, and trained young athletes. The main questions it aims to answer are:

Can EI reliably and accurately measure muscle quality in children when validated against gold-standard techniques like DXA and isokinetic dynamometry? What are the age-, sex-, and fitness-specific benchmarks for EI to differentiate between normal and pathological muscle quality?

ELIGIBILITY:
Inclusion Criteria:

• Generally healthy children

Exclusion Criteria:

* Acute illnesses
* Chronic or acute diseases of the endocrine or musculoskeletal systems
* Post-traumatic conditions

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixty boys and sixty girls aged 10-14 years, evenly distributed as follows: normal-weight children, trained young athletes (≥3 training sessions per week), and obese children according to BMI
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Echo intensity of the vastus lateralis (VL) and rectus femoris (RF) muscles | Through study completion, an average of 1 year
  Echo intensity will be measured by greyscale analysis derivered from ultrasound imaging.

SECONDARY OUTCOMES:
Skeletal Muscle Mass | Through study completion, an average of 1 year
  Measured using DXA (Horizon DXA platform, Hologic)
Muscle Strength | Through study completion, an average of 1 year
  Assessed via isokinetic and isometric knee extensor strength using a Humac Norm isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Sport Charles University, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jandova T, Kinkorova I, Vetrovsky T, Mala J, Musilova E, Steffl M, Narici MV. Can ultrasound echo intensity assess muscle quality in children aged 10-14 years? Protocol for a cross-sectional validation study in Czech children. BMJ Open. 2025 Sep 26;15(9):e100495. doi: 10.1136/bmjopen-2025-100495. PMID 41005786